CLINICAL TRIAL: NCT03196336
Title: Effectiveness of Pharmacotherapy Follow-up Care in Outpatients With Type 2 Diabetes Mellitus: Randomized Clinical Trial
Brief Title: Effectiveness of Pharmacotherapy Follow-up Care in Outpatients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sorocaba (Other)
Collaborators: Cristiane de Cássia Bergamaschi (Unknown)
Responsible Party: Principal Investigator, Luciane Cruz Lopes, PhD, University of Sorocaba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Cristiane
Record Dates: First submitted 2016-10-23; First posted 2017-06-22 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Pharmaceutical Services

STUDY DESIGN:
Intervention Model Description: Pharmacotherapeutic follow-up care known as Pharmacotherapy Workup.
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Other): The intervention is the pharmacotherapeutic follow-up care. This service is performed according to the Pharmacotherapy Workup method, which is a protocol for the pharmacotherapeutic follow-up. This service identify, prevent and solve drug-related problems. It consiste of five pharmaceutical consultations (every up to 2-3 months) with the patient.
  Interventions: Other: Pharmacotherapy follow-up care
- Control (Other): The intervention is the usual procedure of dispensation of drugs. It is performed in five meetings (every up to 2-3 months) between the investigator and the patient.
  Interventions: Other: Pharmacotherapy follow-up care

INTERVENTIONS:
Other: Pharmacotherapy follow-up care — The pharmacotherapy follow-up care consists of five pharmaceutical consultations (every up to 2-3 months) aimed to identify, prevent and solve the drug related problems regarding the indication, effectiveness and safety of the use of medicines.
  Other Names: Pharmacotherapy Workup

SUMMARY:
Hypothesis: Pharmacotherapy follow-up can improve clinical outcomes of outpatients with type 2 diabetes mellitus.

Methods: In this single blind, placebo-controlled trial, the participants with type 2 diabetes mellitus are randomized into two groups:

1. pharmaceutical care intervention (n=30, attended by the protocol of follow-up) and
2. control (n=30, attended by the usual procedure of dispensing).

Primary outcomes evaluated are: hospitalization (percentage of participants hospitalized), severe evolving complication - ischemic or proliferative retinopathy, severe renal insufficiency, severe hypoglycemia, coronaropathy or evolving foot lesion (presence or absence).

Other parameter checked: A1c hemoglobin (HbA1c), blood glucose (BG), blood pressure (BP), total cholesterol (TC), waist circumference (WC), body mass index (BMI) and mortality. The investigators follow up all patients for up to 12 months.

DETAILED DESCRIPTION:
Background. Few Brazilian randomized controlled trials have established the benefits of pharmacotherapy follow-up in care of outpatients with type 2 diabetes mellitus in low-middle income country. This study evaluate the effectiveness of pharmacotherapy follow-up care to get better outcomes in outpatients with type 2 diabetes mellitus attended in the public health service in Brazil.

Method: In this single blind, placebo-controlled trial, the investigators random patients with type 2 diabetes mellitus into two groups: 1) pharmaceutical care intervention (n=30, attended by the protocol of follow-up) and 2) control (n=30, attended by the usual procedure of dispensing).

Primary outcomes checked are: percentage of hospitalization, severe evolving complication (ischemic or proliferative retinopathy, severe renal insufficiency, severe hypoglycemia, coronaropathy and evolving foot lesion).

The investigators also check: A1c hemoglobin (HbA1c), blood glucose (BG), blood pressure (BP), total cholesterol (TC), HbA1c/BP, HbA1c/TC, waist circumference (WC), body mass index (BMI) and mortality. The participants are followed up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

Patients with previous diagnosis of type 2 diabetes, HbA1c greater than 7% and age greater than 18 years

Exclusion Criteria:

Types of diabetes other than type 2 diabetes; patients not responsible for administering their drugs and patients with mental deficits that could no understand the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-03; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
hospitalization | in 12 months
  percentage of participants hospitalized due to diabetes

SECONDARY OUTCOMES:
severe evolving complication (ischemic or proliferative retinopathy, severe renal insufficiency, severe hypoglycemia, coronaropathy or evolving foot lesion) | in 12 months
  number of participants with complication

CONTACTS AND LOCATIONS:
Overall Officials: Cristiane de Cássia Bergamaschi, Principal Investigator — University of Sorocaba
Locations (1):
- Vital Brazil Community Pharmacy, Sorocaba, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
not applied